CLINICAL TRIAL: NCT05097560
Title: The Effect of High Flow Nasal Cannula on Exercise Capacity Compared to Venturi Mask in COPD Patients Recovering From Acute Evacerbation
Brief Title: The Effect of HFNC on Exercise Capacity Compared to VM in COPD Patients Recovering From Acute Evacerbation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Guangzhou Medical University (Other)
Responsible Party: Principal Investigator, Shiying Fang, Principal Investigator, The First Affiliated Hospital of Guangzhou Medical University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FAHGZ-20210811
Record Dates: First submitted 2021-10-16; First posted 2021-10-28 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: COPD
Keywords: HFNC; PR
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HFNC group (Experimental): * Set FiO2 28%
  * Titrate the flow of HFNC at the highest tolerated value up to 60 L/min
  Interventions: Device: high flow nasal cannula
- VM group (Active Comparator): - Keep FiO2 constant with VM and HFNC during the two trial
  Interventions: Device: Venturi mask

INTERVENTIONS:
Device: high flow nasal cannula — HFNC provides humidified, heated, oxygen-enriched air at constant concentration with a flow up to 60L/min through a nasal cannula. It washouts the anatomical dead space and decreases the work of breathing.
  Arms: HFNC group
Device: Venturi mask — VM is commonly used by COPD patients during exercise training.
  Arms: VM group

SUMMARY:
Early PR is thought to be effective in COPD patients recovering from acute exacerbation, while the effect of HFNC during exercise training in these patients remains unclear. The study may provide evidence of early PR in COPD patients recovering from acute exacerbation.

DETAILED DESCRIPTION:
We hypothesize that HFNC may increases exercise time in COPD patients recovering from acute exacerbation compare to VM. A randomized, cross-over clinical trial in which either HFNC or VM may be used as an adjunct in 10-MST in random order, respectively, will be performed to compare the endurance time. The physiological effect of HFNC and VM during exercise will also be measured to explore the mechanism.

ELIGIBILITY:
Inclusion Criteria:

* hospitalized AECOPD patients
* be ambulatory by 48h after admission for AECOPD
* requires oxygen by screening exercise test

Exclusion Criteria:

* active coronary ischemia
* respiratory diseases other than COPD
* unstable vital signs
* unstable psychological status

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2021-08-11 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-08-31 (Estimated)

PRIMARY OUTCOMES:
Endurance time | 10 minute
  Endurance time for 10 minute steping test

SECONDARY OUTCOMES:
Respiratory pattern | 10 minute
  Respiratory pattern is calculated by the flow and time
Work of breathing | 10 minute
  Work of breathing is calculated by the transdiaphragmatic pressure
Neural respiratory drive | 10 minute
  Neural respiratory drive is calculated by diaphragm electromyogram

CONTACTS AND LOCATIONS:
Overall Officials: Rongchang Chen, PhD, Study Chair — The First Affiliated Hospital of Guangzhou Medical University
Locations (1):
- Shiying, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No